CLINICAL TRIAL: NCT02549417
Title: Phase 3 Study of KHK7580 (A Clinical Study of KHK7580 in Subjects With Secondary Hyperparathyroidism Receiving Peritoneal Dialysis)
Brief Title: Phase 3 Study of KHK7580
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7580-012
Record Dates: First submitted 2015-09-09; First posted 2015-09-15 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KHK7580 (Experimental)
  Interventions: Drug: KHK7580

INTERVENTIONS:
Drug: KHK7580 — Oral administration

SUMMARY:
This study is designed to evaluate efficacy and safety of KHK7580 orally administered once daily for 32 weeks for patients with secondary hyperparathyroidism receiving peritoneal dialysis. After 32-week treatment period, the subjects will receive KHK7580 in the 20-week extension period to evaluate long-term safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Personally submitted written voluntary informed consent to participate in the study
* Stable chronic renal disease treated with peritoneal dialysis for at least 16 weeks before screening
* Intact PTH level of > 240 pg/ml at screening

Exclusion Criteria:

* Treatment with cinacalcet hydrochloride within 2 weeks before screening;
* Change in dose or dosing regimen of an activated vitamin D drug or its derivative, phosphate binder, or calcium preparation within 2 weeks before screening; or start of treatment with such drugs within 2 weeks before screening;
* Parathyroidectomy and/or parathyroid intervention within 24 weeks before screening;
* Severe heart disease;
* Severe hepatic dysfunction;
* Uncontrolled hypertension and/or diabetes;
* Treatment with an investigational product (drug or medical device) in a clinical study or any study equivalent to clinical study within 12 weeks before screening;
* Primary hyperparathyroidism;
* Other conditions unfit for participation in this study at the discretion of the investigator or subinvestigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects in the evaluation period achieving a mean intact parathyroid hormone (PTH) level of ≥ 60 pg/mL and ≤ 240 pg/mL | Weeks 30-32

SECONDARY OUTCOMES:
Percentage of subjects in the evaluation period achieving a mean percent decrease in intact PTH level of ≥ 30% (percent change ≤ -30%) from baseline | Weeks 30-32
Mean percent change in the evaluation period in intact PTH level from baseline | Weeks 30-32

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding investigative sites for this trial, contact Kyowa Hakko Kirin, Tokyo, Japan

REFERENCES:
- [Derived] Tsuruya K, Shimazaki R, Fukagawa M, Akizawa T; Evocalcet Study Group. Efficacy and safety of evocalcet in Japanese peritoneal dialysis patients. Clin Exp Nephrol. 2019 Jun;23(6):739-748. doi: 10.1007/s10157-019-01692-y. Epub 2019 Apr 6. PMID 30955188